CLINICAL TRIAL: NCT00911911
Title: Analysis of the Proteomic Signature in Breast Cancer Correlated With Tumor Response in Patients Necessitating a Neo-adjuvant Chemotherapy
Brief Title: Proteomic Signature in Breast Cancer: Correlation With Tumor Response to Neo-adjuvant Chemotherapy
Acronym: SPAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: SPAM 2006-10; NCT00959673 (obsolete NCT alias)
Record Dates: First submitted 2009-05-22; First posted 2009-06-03 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Neo-adjuvant chemotherapy; Proteomic; Histological response
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection; Biopsy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FEC 100 + TAXOTERE (Experimental): FEC 100 = Fluoro-uracile + Epirubicin + Cyclophosphamide Fluoro-uracile : 500 mg/m²/cycle Epirubicin : 100 mg/m²/cycle Cyclophosphamide : 500 mg/m²/cyle 1 cycle = 21 days. For a total of 6 cycles or 3 cycles followed by 3 cycles of TAXOTERE
  TAXOTERE 100 mg/m²/cycle
  1 cycle = 21 days. For a total of 3 cycles following 3 FEC 100
  Interventions: Procedure: Blood sampling; Procedure: BIOPSY; Procedure: SURGERY

INTERVENTIONS:
Procedure: Blood sampling — Taken at different times : inclusion, at the cycle 4 and at the cycle 6 during the neoadjuvant chemotherapy
Procedure: BIOPSY — Biopsy at the moment of inclusion, before neoadjuvant chemotherapy
Procedure: SURGERY — Surgery after neoadjuvant chemotherapy

SUMMARY:
The scope of the trial is to identify proteomic signatures correlated with tumor response to neo-adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Women aged more than 18 years
* Histologically proven breast carcinoma
* Neo-adjuvant chemotherapy with anthracyclines and/or taxanes
* No prior chemotherapy
* Written informed consent

Exclusion Criteria:

* Metastatic disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2007-01; Primary Completion 2009-01 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Proteomic analysis by SELDI-TOF on the tumor biopsy and blood samples Histological response according To Chevallier and Sataloff | 6 months

SECONDARY OUTCOMES:
Correlation with node invasion | 6 months
Correlation with basal, luminal phenotypes, HER2 status or hormonal status | 6 months
Correlation with the response measured by ultrasound after chemotherapy | After 3 and 5 months

CONTACTS AND LOCATIONS:
Overall Officials: BONNETERRE Jacques, MD, PhD, Principal Investigator — Centre Oscar Lambret
Locations (5):
- France (5):
  - Intercommunal Hospital, Annemasse
  - Centre Oscar Lambret, Lille
  - Hopital Saint Vincent, Lille
  - Centre Henri Becquerel, Rouen
  - Geroges PIANTA Hospital, Thonon-les-Bains